CLINICAL TRIAL: NCT04213911
Title: Determination of Pleural Pressure in Subjects With Morbid Obesity
Brief Title: Comparison of Esophageal Manometry and CT Scan Measurements
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Medical doctor, Massachusetts General Hospital
Other Study IDs: CTobese2020
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Morbid Obesity; Respiratory Failure
Keywords: esophageal manometry; superimposed pressure; pleural pressure; chest CT scan
MeSH Terms: conditions — Obesity, Morbid; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morbid obese: BMI>40 kg/m2
  Interventions: Radiation: low-dose chest CT scan; Device: insertion of esophageal balloon
- Non-obese: BMI<30 kg/m2
  Interventions: Radiation: low-dose chest CT scan; Device: insertion of esophageal balloon

INTERVENTIONS:
Radiation: low-dose chest CT scan — The low-dose chest CT scan is now commonly used as a quick, painless, and non-invasive approach to screen for lung cancer. The radiation exposure from one low-dose CT scan of the chest (1.5 mSv) is comparable to 6 months of natural background radiation for a person living in the US.
Device: insertion of esophageal balloon — The esophageal catheter is a flexible thin plastic tube with an air-filled balloon at the distal end. The tube will be placed through the nasopharynx after local anesthesia.

SUMMARY:
The goal of this study is to determine the relationship between esophageal pressure (Pes) and superimposed pressure (SP) in subjects with morbid obesity.

DETAILED DESCRIPTION:
In the clinical setting, Pes is a surrogate for pleural pressure, while SP is measured by means of chest CT scan images. The SP highly approximates the vertical pleural pressure gradient both in normal lungs and injured lungs in lean subjects. It is known that in the healthy obese patient the Pes is higher than that in normal lean patients, but there is no information about the relationship between high Pes with the SP in subjects with morbid obesity.

The investigators hypothesized that factors other than superimposed pressure determine the high Pes in subjects with morbid obesity. Hence, Pes should be high despite the low SP found in healthy obese individuals.

The investigators will test this hypothesis in a prospective observational cohort study.

In 12 subjects (6 with body mass index > 40kg/m2, and 6 with body mass index < 30kg/m2 ) with scheduled chest CT scan for clinical purposes:

1. The Pes will be measured during spontaneous breathing (baseline values at end-expiration and variations during tidal breathing). To achieve this purpose, an esophageal balloon (AVEATM Ventilator Esophageal Pressure Monitoring Tube Set, 8 FR, CareFusion, Yorba Linda, CA, USA) will be inserted after administration of local anesthesia (lidocaine spray 2%).
2. The SP will be determined by lung computed tomography imaging and the pleural pressure will be calculated in non-dependent lung regions as the difference between Pes and SP. For this purpose, an additional low-dose CT scan at the end-expiration will be taken after the scheduled CT scan.

During the research procedure, the Pes during the whole respiratory cycle, the CT image at the end-expiration, demographics, past and current medical history will be recorded.

There will be no follow-up phase in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to take a chest CT scan for the clinical purpose at MGH Radiology Department
* 6 adult subjects with BMI more than 40kg/m2
* 6 adult subjects with BMI less than 30kg/m2
* More than 18 years old

Exclusion Criteria:

* Presence of pneumothorax
* History of spontaneous pneumothorax
* Severe coagulopathy (INR ≥ 4)
* Severe thrombocytopenia (Platelets count ≤ 5,000/mm3)
* Usage of any devices with electric current generation such as pacemakers or internal cardiac defibrillator
* Recent esophageal trauma or surgery
* Other esophageal diseases, such as esophageal cancer, leak, varices, and hernia
* Presence of hypoxemia, short of breath and dysphagia.
* Presence or suspicion of pneumonia or lung fibrosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled to take a chest CT scan without known lung disease. Morbid obesity will be defined as subjects with BMI > 40 kg/m2 and non-obese will be defined as be subjects with BMI < 30 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Esophageal pressure measurement at a given superimposed pressure | through study completion, an average of 1 year
  The esophageal pressure will be determined via esophageal balloon at the end of exhalation. The superimposed pressure will be calculated by chest CT scan image at the end of exhalation.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachussets General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshida T, Amato MBP, Grieco DL, Chen L, Lima CAS, Roldan R, Morais CCA, Gomes S, Costa ELV, Cardoso PFG, Charbonney E, Richard JM, Brochard L, Kavanagh BP. Esophageal Manometry and Regional Transpulmonary Pressure in Lung Injury. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1018-1026. doi: 10.1164/rccm.201709-1806OC. PMID 29323931
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Pelosi P, D'Andrea L, Vitale G, Pesenti A, Gattinoni L. Vertical gradient of regional lung inflation in adult respiratory distress syndrome. Am J Respir Crit Care Med. 1994 Jan;149(1):8-13. doi: 10.1164/ajrccm.149.1.8111603.
- [Background] Hibbert K, Rice M, Malhotra A. Obesity and ARDS. Chest. 2012 Sep;142(3):785-790. doi: 10.1378/chest.12-0117. PMID 22948584
- [Background] Fumagalli J, Berra L, Zhang C, Pirrone M, Santiago RRS, Gomes S, Magni F, Dos Santos GAB, Bennett D, Torsani V, Fisher D, Morais C, Amato MBP, Kacmarek RM. Transpulmonary Pressure Describes Lung Morphology During Decremental Positive End-Expiratory Pressure Trials in Obesity. Crit Care Med. 2017 Aug;45(8):1374-1381. doi: 10.1097/CCM.0000000000002460. PMID 28708679
- [Background] Pirrone M, Fisher D, Chipman D, Imber DA, Corona J, Mietto C, Kacmarek RM, Berra L. Recruitment Maneuvers and Positive End-Expiratory Pressure Titration in Morbidly Obese ICU Patients. Crit Care Med. 2016 Feb;44(2):300-7. doi: 10.1097/CCM.0000000000001387. PMID 26584196
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Mojoli F, Iotti GA, Torriglia F, Pozzi M, Volta CA, Bianzina S, Braschi A, Brochard L. In vivo calibration of esophageal pressure in the mechanically ventilated patient makes measurements reliable. Crit Care. 2016 Apr 11;20:98. doi: 10.1186/s13054-016-1278-5. PMID 27063290
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] American College of Radiology and Radiological Society of North America. https://www.radiologyinfo.org/en/info.cfm?pg=safety-xray.
- [Background] National Cancer Institute at the National Institutes of Health. Computed Tomography (CT): Questions and Answers. [July 20, 2012]; Available from: http:://www.cancer.gov/cancertopics/factsheet/detection/CT.